CLINICAL TRIAL: NCT04048486
Title: Follow-up of Children Born From CAPA-IVM IVF or Natural Conception: a Prospective Cohort Study
Brief Title: Children Born From IVM-CAPA vs IVF or Natural Conception
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CS/BVMĐ/19/07
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: IVM; IVF
MeSH Terms: interventions — Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CAPA-IVM: Live babies born from CAPA-IVM
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags
- IVF/ICSI: Live babies born from IVF/ICSI
- Natural conception: Live babies born from natural conception
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags

INTERVENTIONS:
Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy-to-use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones.
  Groups: CAPA-IVM; Natural conception
Other: Physical development and General Health — Physical development and General health examination
  Groups: CAPA-IVM; Natural conception
Other: Developmental Red flags — Developmental Red flags Questionnaires
  Groups: CAPA-IVM; Natural conception

SUMMARY:
CAPA-IVM is a new promising IVM technique involving the use of a new compound to facilitate the oocyte and embryo competence. CAPA-IVM preserved the maintenance of trans-zonal projections and significantly improved maturation rate and blastocyst yield. NGS analysis of 20 good quality CAPA-IVM blastocysts did not reveal increased aneuploidy compared to age-matched routine ICSI patients. The first CAPA-IVM baby was born in 2017 at My Duc Hospital, Vietnam and up to now, there are 33 babies born from this technique. There is no study to investigate the development of babies born from CAPA-IVM.

DETAILED DESCRIPTION:
Assisted reproductive technologies (ART), such as in vitro fertilization (IVF), intracytoplasmic sperm injection (ICSI) and in vitro maturation (IVM), are widely used to solve human infertility, and have provided great benefits for millions of couples who have struggled with infertility disorders. The use of ART has been growing persistently and more than 8 million babies worldwide have been born via ART since the first IVF conceived child was born in 1978 (ESHRE monitoring).

During the last two decades, many studies have shown that children born following assisted reproductive techniques (ART) have an increased risk of adverse obstetric, perinatal and short-term follow-up outcomes when compared to naturally conceived (NC) infants (Jackson RA 2004, Helmerhorst et al., 2004; Pinborg et al., 2013; Adams et al., 2015). The etiologies of this association are mainly related to higher proportion of multiple pregnancies due to double embryo transfer option and greater rate of unfavorable comorbidities of infertile women (older age, high BMI, diabetes…). But with the trend toward single embryo transfer in current IVF practice, there are existing evidences supporting that the perinatal risks of singleton gestations following IVF treatment are still higher than those that result from a spontaneous conception (McDonald et al., 2009; Pandey et al., 2012).

Long-term development of children born by ART is also a concerned issue. It is evident that children born as a result of IVF treatment have an excess rate of congenital abnormalities, higher risk of developing metabolic, cardiovascular disorders and subclinical hyperthyroidism in later life (Roger Hart and Robert J. Norman, 2013, part I). Regarding mental health and development outcomes, cerebral palsy and slight neurodevelopmental delay are potential long-term associations with ART (Roger Hart and Robert J. Norman, 2013, part II). However, these adverse outcomes can be explained by obstetric factors (higher rate of prematurity and intrauterine growth restriction) rather than IVF. This leads to the concern about research biases in studies of long-term development of children born by ART where multiple gestations, prematurity, neonatal hospitalization and growth restriction were not well-controlled. Another concern about long-term follow-up studies of IVF children is the limitation of literatures and high-quality clinical trials that investigate the general health outcomes of children born by ART. The majority of valuable data only exist on the short-term outcome of infants born as a result of IVF treatment (Kalra and Barnhart, 2011) even though it is possible that some suspected disorders might only be identifiable beyond the first year of life (Oliver et al., 2012).

When studying about the long-term development of children following ART, a very important factor need to be considered is the medium of culture. There have been existing theories that proposed the mechanism of how epigenetic environment can up or down-regulate a set of genes which then results in the changes in embryonic growth or even the long-term development of children in later stage of life. Different ART methods may cause possible changes in DNA methylation patterns which in turn affect development of the placenta and fetus. This is the "developmental origins of health and disease hypothesis" (DOHaD) explaning why exposure to an adverse environment (possibly the culture medium) may result in unfavorable development and illnesses profiles in the ART offspring (Barker, 2007).

CAPA-IVM is a new promising IVM technique involving the use of a new compound to facilitate the oocyte and embryo competence. CAPA-IVM preserved the maintenance of trans-zonal projections and significantly improved maturation rate and blastocyst yield. NGS analysis of 20 good quality CAPA-IVM blastocysts did not reveal increased aneuploidy compared to age matched routine ICSI patients. The first CAPA-IVM baby was born in 2017 at My Duc Hospital, Vietnam and up to now, there are 33 babies born from this technique. There is no study to investigate the development of babies born from CAPA-IVM.

The investigators therefore conduct this study to investigate the physical and mental development of babies born from CAPA-IVM, IVF or natural conception.

ELIGIBILITY:
Inclusion Criteria:

* Live babies born from CAPA-IVM
* Live babies born from IVF
* Live babies born from natural conception
* Parents agree to participate

Exclusion Criteria:

* Babies born from oocyte donation cycles
* Babies born from sperm donation cycles
* Babies born from PGT cycles

Ages: 1 Month to 66 Months | Sex: All
Age Groups: Child
Study Population: Live babies born from CAPA-IVM, IVF or natural conception
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
The average total ASQ-3 score | Up to 66 months after birth
  * ASQ-3 (Ages and Stages Questionares®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social
  * Each aspesct has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  * ASQ-3 average = average score of 5 aspects.

SECONDARY OUTCOMES:
Score of Communication | Up to 66 months after birth
  * 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  * Total score will be used: minimum = 0 and maximum = 60.
  * Each aspects in each stages has alternative threshold
Score of Gross motor | Up to 66 months after birth
  * 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  * Total score will be used: minimum = 0 and maximum = 60.
  * Each aspects in each stages has alternative threshold
Score of Fine motor | Up to 66 months after birth
  * 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  * Total score will be used: minimum = 0 and maximum = 60.
  * Each aspects in each stages has alternative threshold
Score of Problem solving | Up to 66 months after birth
  * 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  * Total score will be used: minimum = 0 and maximum = 60.
  * Each aspects in each stages has alternative threshold
Score of Personal-Social | Up to 66 months after birth
  * 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  * Total score will be used: minimum = 0 and maximum = 60.
  * Each aspects in each stages has alternative threshold
The presence of red flag signs by age | Up to 24 months after birth
  1. For children less than 4 months
     * Rolling prior to 3 months
     * Persistent fisting at 3 months
     * Failure to alert to environmental stimuli
  2. For children from 4 to 6 months
     * Poor head control
     * Failure to reach for objects by 5 months
     * Absent smile
  3. For children from 6 to 12 months
     * Absent babbling by 6 months
     * W-sitting at 7 months
     * Inability to localize sound by 10 months
     * Persistent mouthing of objects at 12 months
     * Lack of consonant production by 15 months
  4. For children from 12 to 24 months
     * Lack of imitation by 16 months
     * Lack of protodeclarative pointing by 18 months
     * Hand dominance prior to 18 months
     * Inability to walk up and down stairs at 24 months
     * Advanced non-communicative speech (meaningless communication repertoires)
     * Delayed Language Development milestone (50 single words at 24 months)
Duration of breast-feeding | Up to 24 months after birth
  Duration of breast-feeding
Infant age at which weaning starts | Up to 24 months after birth
  Infant age at which weaning starts
Diseases that lead to hospital admission | Up to 24 months after birth
  Diseases that lead to hospital admission
Number of hospital admission | Up to 24 months after birth
  Number of hospital admission
Weight | At 3, 6, 12, 18, 24 months and on the examination date
  Weight at 3, 6, 12, 18, 24 months and on the examination date
Height | At 3, 6, 12, 18, 24 months and on the examination date
  Height at 3, 6, 12, 18, 24 months and on the examination date

OTHER OUTCOMES:
Gestational age at delivery | At birth
  Gestational age at delivery
Mode of delivery | At birth
  Vaginal birth or C-section
Birth weight | At birth
  Weight of baby born
Length circumference | At birth
  Length circumference after birth
Head circumference | At birth
  Head circumference after birth
Rate of congenital anomalies | At birth
  Any congenital anomalies detected in baby born
5-min Apgar score | At 5 minute after birth
  The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration).
Rate of 5-min Apgar score <7 | At 5 minute after birth
  Rate of Apgar score at 5 minute after birth <7
Rate of Admission to neonatal intensive care unit | Within 7 days after birth
  Admission to neonatal intensive care unit of baby
Length of NICU admission | Up to 28 days after birth
  Number of admission days to NICU
Rate of Respiratory distress syndrome | Up to 28 days after birth
  Respiratory distress syndrome (RDS), diagnosed as the presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram.
Rate of Periventricular haemorrhage | Up to 28 days after birth
  Periventricular haemorrhage II B or worse, will be diagnosed by repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al.
Rate of Necrotizing enterocolitis | Up to 28 days after birth
  Necrotizing enterocolitis (NEC) will be diagnosed according to Bell.
Rate of Proven sepsis | Up to 28 days after birth
  Proven sepsis, will be diagnosed on the combination of clinical signs and positive blood cultures.
Rate of Composite of poor perinatal outcomes | Up to 28 days after birth
  Composite of poor perinatal outcomes, defined as intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stephens SM, Arnett DM, Meacham RB. The use of in vitro fertilization in the management of male infertility: what the urologist needs to know. Rev Urol. 2013;15(4):154-60. PMID 24659912
- [Background] Helmerhorst FM, Perquin DA, Donker D, Keirse MJ. Perinatal outcome of singletons and twins after assisted conception: a systematic review of controlled studies. BMJ. 2004 Jan 31;328(7434):261. doi: 10.1136/bmj.37957.560278.EE. Epub 2004 Jan 23. PMID 14742347
- [Background] Pinborg A, Wennerholm UB, Romundstad LB, Loft A, Aittomaki K, Soderstrom-Anttila V, Nygren KG, Hazekamp J, Bergh C. Why do singletons conceived after assisted reproduction technology have adverse perinatal outcome? Systematic review and meta-analysis. Hum Reprod Update. 2013 Mar-Apr;19(2):87-104. doi: 10.1093/humupd/dms044. Epub 2012 Nov 14. PMID 23154145
- [Background] McDonald SD, Han Z, Mulla S, Murphy KE, Beyene J, Ohlsson A; Knowledge Synthesis Group. Preterm birth and low birth weight among in vitro fertilization singletons: a systematic review and meta-analyses. Eur J Obstet Gynecol Reprod Biol. 2009 Oct;146(2):138-48. doi: 10.1016/j.ejogrb.2009.05.035. Epub 2009 Jul 4. PMID 19577836
- [Background] Pandey S, Shetty A, Hamilton M, Bhattacharya S, Maheshwari A. Obstetric and perinatal outcomes in singleton pregnancies resulting from IVF/ICSI: a systematic review and meta-analysis. Hum Reprod Update. 2012 Sep-Oct;18(5):485-503. doi: 10.1093/humupd/dms018. Epub 2012 May 19. PMID 22611174
- [Background] Hart R, Norman RJ. The longer-term health outcomes for children born as a result of IVF treatment: Part I--General health outcomes. Hum Reprod Update. 2013 May-Jun;19(3):232-43. doi: 10.1093/humupd/dms062. Epub 2013 Feb 28. PMID 23449642
- [Background] Hart R, Norman RJ. The longer-term health outcomes for children born as a result of IVF treatment. Part II--Mental health and development outcomes. Hum Reprod Update. 2013 May-Jun;19(3):244-50. doi: 10.1093/humupd/dmt002. Epub 2013 Feb 28. PMID 23449643
- [Background] Kalra SK, Barnhart KT. In vitro fertilization and adverse childhood outcomes: what we know, where we are going, and how we will get there. A glimpse into what lies behind and beckons ahead. Fertil Steril. 2011 May;95(6):1887-9. doi: 10.1016/j.fertnstert.2011.02.044. Epub 2011 Mar 16. PMID 21411083
- [Background] Oliver VF, Miles HL, Cutfield WS, Hofman PL, Ludgate JL, Morison IM. Defects in imprinting and genome-wide DNA methylation are not common in the in vitro fertilization population. Fertil Steril. 2012 Jan;97(1):147-53.e7. doi: 10.1016/j.fertnstert.2011.10.027. Epub 2011 Nov 23. PMID 22112648
- [Background] Barker DJ. The origins of the developmental origins theory. J Intern Med. 2007 May;261(5):412-7. doi: 10.1111/j.1365-2796.2007.01809.x. PMID 17444880
- See also: De Geyter — https://www.eshre.eu/Annual-Meeting/Barcelona-2018/ESHRE-2018-Press-releases/De-Geyter
- See also: Adams: A meta-analysis of neonatal health outcomes — https://scholar.google.com/scholar_lookup?title=A%20meta-analysis%20of%20neonatal%20health%20outcomes%20from%20oocyte%20donation&author=D%20Adams&author=R%20Clark&author=M%20Davies&author=S%20De%20Lacey&publication_year=2016&journal=J%20Dev%20Orig%20Health%20Dis&volume=7&pages=257-272